CLINICAL TRIAL: NCT01026792
Title: A Phase II Study of Temsirolimus (NSC 683864), an mTOR Inhibitor, in Patients With Recurrent, Unresectable, Locally Advanced or Metastatic Carcinoma of the Cervix
Brief Title: Temsirolimus in Treating Patients With Cervical Cancer That Is Recurrent, Locally Advanced, Metastatic, or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00268; NCI-2014-00268 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCIC-CTG-199; CDR0000660702; IND.199; CAN-NCIC-IND199; NCIC-199 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-199 (Other: CTEP)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma; Stage IIIA Cervical Cancer; Stage IIIB Cervical Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. For complete responders, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity or for 2 courses after complete response criteria are first met. For other patients, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Temsirolimus; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; Torisel
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the effects of temsirolimus in treating patients with cervical cancer that cannot be cured by standard therapy. Temsirolimus interferes with a protein in cells that is part of one pathway that sends signals to stimulate cell growth and survival. By blocking this protein cancer cells may stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (objective response rate) of temsirolimus given intravenously (IV) weekly in patients with metastatic and/or locally advanced recurrent carcinoma of the cervix.

II. To assess the adverse events, time to progression and response duration of temsirolimus given IV weekly in patients with metastatic and/or locally advanced recurrent carcinoma of the cervix.

III. To explore the relationship between expression of proteins in the mammalian target of rapamycin (mTOR) pathway in archival tissue samples from patients on this trial and their objective response to therapy.

OUTLINE:

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. For complete responders, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity or for 2 courses after complete response criteria are first met. For other patients, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months (patients with complete response [CR], partial response [PR], or stable disease [SD] only) thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell carcinoma or adenosquamous carcinoma of the cervix, or adenocarcinoma of the cervix
* Patients must have unresectable, locally advanced or metastatic disease, incurable by standard therapies
* Patients must have tumor tissue from their primary tumor available
* Presence of clinically and/or radiologically documented disease

  * Chest x-ray >= 20 mm
  * Computed tomography (CT) scan (with slice thickness of =< 5 mm) >= 10 mm: longest diameter
  * Physical exam (using calipers) >= 10 mm
  * Lymph nodes by CT scan >= 15 mm: measured in short axis
  * All radiology studies must be performed within 21 days prior to registration (within 28 days if negative)
* Patients must have a life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients may have had up to one prior chemotherapy regimen; a minimum of 28 days (4 weeks) must have elapsed between the end of chemotherapy and study registration; Note: Radiotherapy with concurrent radiosensitizing cisplatin at the time of initial diagnosis and treatment is permitted, and is not considered systemic chemotherapy
* Patients may have had prior radiation therapy; a minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study; (exceptions may be made however, for low dose, palliative radiotherapy); patients must have recovered from any acute toxic effects from radiation prior to registration
* Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred
* Granulocytes (AGC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Serum creatinine =< 1.5 upper limit of normal (ULN)
* Bilirubin =< 1.5 ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Fasting serum cholesterol =< 9.0 mmol/L
* Fasting triglycerides =< 2.5 x ULN
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements; it will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the National Cancer Institute of Canada (NCIC) Clinical Trials Group (CTG) study coordinator that such clearance has been obtained, before the trial can commence in that center; a standard consent form for the trial will not be provided but a sample form is given; a copy of the initial full board Research Ethics Board (REB) approval and approved consent form must be sent to the central office; the patient must sign the consent form prior to registration; please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records
* Patients must be accessible for treatment, response assessment and follow-up; patients registered on this trial must be treated and followed at the participating center; this implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial; investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for >= 5 years
* Patients must not have had prior treatment with an mTOR inhibitor
* Pregnant or lactating women; pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with temsirolimus; if the patient is of childbearing potential, a urine beta (β)-human chorionic gonadotropin (HCG) must be proved negative within 7 days prior to registration; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with known brain metastases (a brain CT is not necessary to rule out brain metastases, unless there is clinical suspicion of CNS involvement); patients with known brain metastases will be excluded from this trial
* Patients with serious cardiovascular illness such as myocardial infarction within 6 months prior to entry, congestive heart failure (even if medically controlled), unstable angina, active cardiomyopathy, unstable ventricular arrhythmia or uncontrolled hypertension
* Patients who require use of therapeutic anticoagulation are ELIGIBLE but must have their prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) monitored closely during therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational agents
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements
  * Active uncontrolled infection or non-healing wounds
  * Active peptic ulcer disease
  * Active bleeding or any other medical conditions that might be aggravated by treatment
  * Symptomatic congestive heart failure, unstable angina, cardiac arrhythmia
  * Fistula or history of fistula at any location, gastrointestinal (GI) perforation or abscess; patients believed to be at high risk for fistula formation because of the location and extent of their disease should not be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tinker, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Temsirolimus)
Started | 38
Completed | 37
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 50 [26 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Response is defined as a 30% decrease in the sum of the longest diameters of the target lesions (PR) or complete disappearance of disease and symptoms (CR) for at least 4 weeks as assessed by Response Evaluation Criteria in Solid Tumors 1.1
Time Frame: Up to 3 years
Population: Patients evaluable for response
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 33
percentage of patients with response | 3 [0.1 to 15.8]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 15/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=37)
Edema: limb (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Death NOS (General disorders) | 6
Hematuria (Renal and urinary disorders) | 2
Paresthesia (Nervous system disorders) | 1
Other renal and urinary disorders (Renal and urinary disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=37)
Anemia (Blood and lymphatic system disorders) | 5
Palpitations (Cardiac disorders) | 2
Other ear and labyrinth disorders (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 10
Bloating (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 20
Rectal hemorrhage (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 12
Other gastrointestinal disorders (Gastrointestinal disorders) | 13
Chills (General disorders) | 4
Edema face (General disorders) | 3
Edema limbs (General disorders) | 15
Fatigue (General disorders) | 30
Fever (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 9
Other general disorders, administration site conditions (General disorders) | 2
Urinary tract infection (Infections and infestations) | 7
Other infections and infestations (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 4
Weight gain (Investigations) | 3
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 18
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 13
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 18
Hematuria (Renal and urinary disorders) | 5
Urinary frequency (Renal and urinary disorders) | 7
Urinary tract obstruction (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 4
Urinary urgency (Renal and urinary disorders) | 2
Other renal and urinary disorders (Renal and urinary disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 5
Vaginal discharge (Reproductive system and breast disorders) | 5
Vaginal hemorrhage (Reproductive system and breast disorders) | 4
Other reproductive system and breast disorders (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Lymphedema (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less